CLINICAL TRIAL: NCT03304002
Title: Implementation of a Web-based Decision Aid for Breast Cancer Surgery: Adapting to the Needs of Diverse Settings
Brief Title: Implementation of a Web-based Decision Aid for Breast Cancer Surgery
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2017-0588; A539740 (Other: UW Madison); SMPH\SURGERY\GEN SURG (Other: UW Madison); 5P30CA014520-43 (NIH); UW16147 (Other: UWCCC); Protocol Version 3/15/2019 (Other: UW Madison)
Record Dates: First submitted 2017-09-27; First posted 2017-10-06 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Breast Cancer; Surgery
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Breast Cancer Surgery Decision Aid — We use a standard decision aid collaboratively developed by Health Dialog and the Informed Medical Decisions Foundation

SUMMARY:
Routine incorporation of decision aids into oncology practice has the potential to significantly improve patients' experiences with cancer by increasing the likelihood that they make informed treatment decisions aligned with their values. Unfortunately, only a minority of the more than 1.6 million patients diagnosed annually with cancer ever receive one due to limited clinic resources for administration and challenges in timely identification of appropriate patients. Online delivery directly to patients addresses some of these barriers but is insufficient on its own to ensure accessibility for patients at the time they most benefit from support.19 It is critical that active, multi-faceted implementation strategies that target barriers to the widespread use of web-based decision aids be identified, as these tools have the potential to significantly improve the quality of oncologic care.

Based on strong preliminary work, the investigators have developed and piloted a package of implementation strategies that effectively overcomes barriers to delivery of a web-based breast cancer surgery decision aid in an academic and community clinic. Although the strategy was successful, patients were white and educated; further investigation is imperative in settings that provide care to underserved patients to ensure the intervention will mitigate, rather than worsen, existing disparities in breast cancer care. This is especially critical given that underserved patients may benefit most from shared decision-making interventions such as the one described. To study this, the investigators propose a pilot study within a clinic that serves a catchment area with a high proportion of African American, rural and low income patients. The investigators will iteratively assess and enhance our implementation package using concepts outlined in the Knowledge-to-Action Cycle, which emphasizes local context in balancing fidelity and flexibility. The specific aims are: 1) To identify patient and clinic level barriers to implementation of a web-based breast cancer surgery decision aid in a clinic that cares for underserved patients, and 2) To test and expand our current implementation package's ability to address barriers in a clinic that cares for underserved patients. The investigators will determine the reach of implementation and acceptability of this method of decision aid delivery to stakeholders.

ELIGIBILITY:
Patients:

Inclusion Criteria:

* Patients newly diagnosed with Stage 0-3 breast cancer.

Exclusion Criteria:

* None

Clinic Stakeholders:

Inclusion Criteria: clinical staff, clinic leadership, and surgeons involved in implementation Exclusion Criteria: none

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a clinic-level intervention with two stakeholder groups: (1) clinical staff, clinic leadership, and surgeons involved in implementation, and (2) patients newly diagnosed with Stage 0-3 breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2020-05-12 (Actual); Study Completion 2020-05-12 (Actual)

PRIMARY OUTCOMES:
Reach: Proportion of Participants who Utilize the Decision Aid | measured over the 4 month implementation period
  Reach of the implementation is defined as the proportion of participants over the four month implementation period who: 1) are sent the decision aid and 2) access the decision aid.

SECONDARY OUTCOMES:
Acceptability: Percentage of Participants Who Would Recommend Receiving Breast Cancer Information Via Email | Survey sent within 4 weeks of surgical consultation
  acceptability will be defined as >80% of patients reporting they would recommend receiving breast cancer information via email to others.
Barriers and Facilitators to Implementation of the Decision Aid | Interviewed completed within 6 months of the surgical consultation
  One-on-one interviews with participants to identify those who experienced barriers and facilitators to implementing the decision aid

CONTACTS AND LOCATIONS:
Overall Officials: Heather Neuman, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - Baptist Health System, Memphis, Tennessee
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin